CLINICAL TRIAL: NCT03643289
Title: Predicting Response to Immunotherapy for Melanoma With Gut Microbiome and Metabolomics
Acronym: PRIMM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: RD2016-56
Record Dates: First submitted 2018-08-10; First posted 2018-08-22 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples, blood samples, tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Patients with stage 4 melanoma due to commence immunotherapy. Patients should be naïve to immunotherapy.
- Cohort B: Patients with stage 3 melanoma who are naïve to immunotherapy

SUMMARY:
This study will investigate the effects of gut microbiome diversity (richness in terms of many bacterial species in the gut) on responses and side effects of immunotherapy in advanced melanoma patients. Immunotherapy for melanoma is especially damaging for the gut with colitis which can lead to death and significant morbidity with repeated hospital admissions. The richness of the microbiome in the gut may be protective against colitis and other side effects but this needs to be confirmed. There is also some preliminary evidence that the gut microbiome diversity can enhance responses to immunotherapy in cancer but this has been shown in small numbers of melanoma patients.

DETAILED DESCRIPTION:
This pilot project will assess the gut microbiome with metagenome sequencing before and after starting immunotherapy in stage 3 and 4 melanoma patients. The project will assess the impact of the gut microbiome on treatment response rates and side effects induced by immunotherapy.

200 stage 4 and 250 stage 3 melanoma patients naive to immunotherapy will be recruited from melanoma clinics. Stool samples will be donated pre-treatment and at follow-up visits throughout treatment. An additional sample will also be requested in the event of disease progression or toxicity necessitating treatment delay or discontinuation. An accompanying stool sample questionnaire will be completed at each sampling time point with the optional completion of a 24-hour recall food diary.

Blood samples will also be taken before and after starting immunotherapy treatment, with gastrointestinal, food frequency, quality of life questionnaires administered at baseline. An optional tumour biopsy if safe and accessible, is requested from patients in the stage 4 cohort before and after starting immunotherapy.

Microbiome data from melanoma patients will be compared with the TwinsUK healthy control gut microbiome data on more than 3000 healthy adults. This analysis will help us assess if there are major differences between the microbiome composition in the melanoma cases prior to therapy compared to the control gut microbiome data from TwinsUK.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged over the age of 18 years with advanced melanoma due to receive first line systemic treatment with immunotherapy with a checkpoint inhibitor alone or in combination.

Exclusion Criteria:

* Patients who have had systemic anti-cancer treatment for locally advanced or metastatic disease.
* Patients unable to consent because of language barrier or inability to consent.
* Patients unable to collect or send the stool samples for geographical, social or psychological reasons.
* Persons benefitting from protection system of adults (including guardianship and curatorship)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 3 or 4 melanoma
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2023-05-02 (Estimated); Study Completion 2023-05-02 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome diversity via measurement of bacterial species in stool samples | 3-5 years
  Gut microbiome diversity and peripheral blood mononuclear cells immunophenotyping in relation to responses to treatment and side effects in patients with stage 3 or stage 4 melanoma receiving immunotherapy
Peripheral blood monocyte measurements to determine the characterisation of peripheral blood mononuclear cells (immunophenotyping) and inflammatory markers before and after starting immunotherapy treatment. | 3-5 years
  Gut microbiome diversity and peripheral blood mononuclear cells immunophenotyping in relation to responses to treatment and side effects in patients with stage 3 or stage 4 melanoma receiving immunotherapy.
Side effects as determined by CTCAE scale Common Toxicity Criteria for Adverse Events v5.03 | 3-5 years
  Gut microbiome diversity and peripheral blood mononuclear cells immunophenotyping in relation to responses to treatment and side effects in patients with stage 3 or stage 4 melanoma receiving immunotherapy.

SECONDARY OUTCOMES:
Analysis of optional punch biopsy samples before and after commencing immunotherapy treatment in patients with stage 4 melanoma | 3-5 years
  Exploratory analysis to examine the association between the gut microbiome and the presence of tumour infiltrates and regulatory environments.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston

IPD SHARING:
Plan to Share IPD: No
The research results will be published in international journals and presented at scientific meetings.